CLINICAL TRIAL: NCT03199300
Title: Investigating Cardiovascular Adverse Events Related to Cancer Treatment: a Study of Extreme Toxicity Using Induced Pluripotent Stem Cells
Brief Title: Investigating Cardiovascular Adverse Events Related to Cancer Treatment
Acronym: InvestiCAT
Status: Active, not recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: 201700454
Record Dates: First submitted 2017-06-22; First posted 2017-06-26 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Toxicity Due to Chemotherapy; Cardiovascular Morbidity; Cancer, Treatment-Related
Keywords: bleomycin; cisplatin; trastuzumab; anthracyclines; toxicity
MeSH Terms: conditions — Neoplasms, Second Primary | interventions — Anthracyclines; Trastuzumab; Cisplatin; Bleomycin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Urine sample, blood sample, germline DNA, skin fibroblasts.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Anthracylines-treated with toxicity: Patients with toxicity during/after treatment with anthracylines.
  Interventions: Drug: Anthracyclines
- Anthracyclines-treated without toxicity: Patients without toxicity during/after treatment with anthracylines.
  Interventions: Drug: Anthracyclines
- Trastuzumab-treated with toxicity: Patients with toxicity during/after treatment with trastuzumab.
  Interventions: Drug: Trastuzumab
- Trastuzumab-treated without toxicity: Patients without toxicity during/after treatment with trastuzumab.
  Interventions: Drug: Trastuzumab
- Cisplatin-treated with toxicity: Patients with toxicity during/after treatment with cisplatin.
  Interventions: Drug: Cisplatin
- Cisplatin-treated without toxicity: Patients without toxicity during/after treatment with cisplatin.
  Interventions: Drug: Cisplatin
- Bleomycin-treated with toxicity: Patients with toxicity during/after treatment with bleomycin.
  Interventions: Drug: Bleomycin
- Bleomycin-treated without toxicity: Patients without toxicity during/after treatment with bleomycin.
  Interventions: Drug: Bleomycin

INTERVENTIONS:
Drug: Anthracyclines — Chemotherapy regimen containing anthracyclines.
  Groups: Anthracyclines-treated without toxicity; Anthracylines-treated with toxicity
Drug: Trastuzumab — Systemic treatment including trastuzumab.
  Groups: Trastuzumab-treated with toxicity; Trastuzumab-treated without toxicity
Drug: Cisplatin — Chemotherapy including cisplatin.
  Groups: Cisplatin-treated with toxicity; Cisplatin-treated without toxicity
Drug: Bleomycin — Chemotherapy including bleomycin.
  Groups: Bleomycin-treated with toxicity; Bleomycin-treated without toxicity

SUMMARY:
Cisplatin, anthracyclines, bleomycin and trastuzumab can cause severe cardiovascular or pulmonary toxicity. Why some patients are susceptible to extreme toxicity of cancer treatment is largely unknown. Unraveling extreme cardiovascular toxic responses in cancer patients may help understand the pathophysiology of cardiovascular toxicity of these agents and help in understanding the more subtle, long-term cardiovascular side effects that affect a larger part of cancer survivors. With induced pluripotent stem cells we will obtain patient-derived cells to recapitulate and mimic and study pathological (cardiovascular) responses and (cardiovascular) toxicity in vitro.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of these criteria:

1. any proven cancer treated with curative intent;
2. age ≥ 18 and ≤ 50 years;
3. able to comply with the protocol;
4. signed written informed consent.

There are specific inclusion criteria for every subject group:

* severe toxicity during 1 to 3 cycles of anthracyclines;
* ≥ 3 months after end of cancer treatment which included the maximum tolerable dose of anthracyclines without (severe) toxicity;
* severe toxicity within 1 to 6 cycles of trastuzumab;
* ≥ 3 months after end of cancer treatment which included a year of trastuzumab without (severe) toxicity.
* severe toxicity during 1 to 3 cycles of cisplatin;
* ≥ 1 year after end of cancer treatment which included high-dose cisplatin without toxicity;
* severe toxicity during 1 to 3 cycles of bleomycin;
* ≥ 1 year after end of cancer treatment which included high-dose bleomycin without toxicity.

Severe toxicity is defined as any of grade 3 - 4 toxicity according to CTCAE 4.03.

A potential subject who meets any of the following exclusion criteria will be excluded from participation in this study:

1. history of cardiovascular disease prior to start of cancer treatment, as evidenced by any of the following: symptomatic or treated cardiovascular disease prior to start of cancer treatment; LVEF < 55% at any performed MUGA scan or echocardiography prior to start of cancer treatment;
2. any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol, or insufficient understanding of the Dutch language;
3. any contraindication for skin biopsy, including: extensive skin disorder precluding biopsy of unaffected skin; known allergy to local anaesthetics; use of anticoagulants and INR > 3;
4. pregnant or lactating female.

   Furthermore, there are specific exclusion criteria for the control groups:
5. history of cardiovascular disease during or after cancer treatment, as evidenced by any of the following: any symptomatic or treated cardiovascular disease; LVEF < 55% at any performed MUGA scan or echocardiography.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated for a malignancy with any of the described cytotoxic agents.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2025-02-06 (Actual); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Comparison between iPSC-derived cells | 3 years
  Comparison between iPSC-derived cells from toxicity cases and controls, for each of the four different agents.

SECONDARY OUTCOMES:
Correlate the findings from the iPSC-derived cells with the clinical phenotype of cardiovascular toxicity | 3 years
  Correlate the findings from the iPSC-derived cells with the clinical phenotype of (cardiovascular) toxicity, assessed by circulating biomarkers and cardiac or vascular imaging.

CONTACTS AND LOCATIONS:
Overall Officials: J.A. Gietema, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No